CLINICAL TRIAL: NCT02571283
Title: A Randomized, Prospective Trial Comparing Peri-articular Injection Utilizing a Pain Cocktail With and Without Exparel
Brief Title: Peri-articular Injection Utilizing a Pain Cocktail With and Without Exparel
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI decided to focus on more current topics of interest.
Sponsor: University of Louisville (Other)
Collaborators: Arthroplasty Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14.1276
Record Dates: First submitted 2015-09-28; First posted 2015-10-08 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Total Knee Arthroplasty; Pain Management
Keywords: Total Knee Arthroplasty; Total Knee Replacement; Exparel; Cocktail Injection; Pain Management
MeSH Terms: conditions — Agnosia | interventions — Ropivacaine; Ketorolac Tromethamine; Ketorolac; Epinephrine; Clonidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Randomized Group A [Cocktail Injection] (Experimental): COCKTAIL INJECTION:
  Cocktail Injection Consists of:
  Ropivacaine (Brand Name: Naropin) 5 mg/ml (49.25 ml) Ketorolac (Brand Names: Toradol, Sprix, Acuvail, Acular) 30 mg/ml (1 ml) Epinephrine (Brand Names: EpiPen, Adrenaclick, Medihaler-Epi, Twinject) 1 mg/ml (0.5 ml) Clonidine (Brand Names: Kapvay, Catapres, Duraclon, Nexiclon) 0.1 mg/ml (0.08 mg = 0.8 ml) Normal Saline added to total of 100 cc Dosage Form: Injection Dosage: See above Frequency: Single dose
  Interventions: Drug: Cocktail
- Randomized Group B [Cocktail Injection Plus Exparel] (Experimental): COCKTAIL INJECTION PLUS EXPAREL:
  Cocktail Injection Consists of:
  Ropivacaine (Brand Name: Naropin) 5 mg/ml (49.25 ml) Ketorolac (Brand Names: Toradol, Sprix, Acuvail, Acular) 30 mg/ml (1 ml) Epinephrine (Brand Names: EpiPen, Adrenaclick, Medihaler-Epi, Twinject) 1 mg/ml (0.5 ml) Clonidine (Brand Names: Kapvay, Catapres, Duraclon, Nexiclon) 0.1mg/ml (0.08 mg = 0.8 ml) Normal Saline added to total of 100 cc Dosage Form: Injection Dosage: See above Frequency: Single dose
  Bupivacaine Liposome (Brand Name: Exparel) Dosage Form: Injection Dosage: 20 ml Single use vial, 1.3% (13.3 mg/ml) Frequency: Single dose
  Interventions: Drug: Cocktail; Drug: Exparel
- Randomized Group C [Marcaine Plus Exparel] (Experimental): MARCAINE PLUS EXPAREL:
  Bupivacaine Hydrochloride (Brand Name: Marcaine, Sensorcaine) Dosage Form: Injection Dosage: 3 ml vial, 0.5% solution Frequency: Single dose
  Bupivacaine Liposome (Brand Name: Exparel) Dosage Form: Injection Dosage: 20 ml Single use vial, 1.3% (13.3 mg/ml) Frequency: Single dose
  Interventions: Drug: Exparel; Drug: Marcaine

INTERVENTIONS:
Drug: Cocktail — Administered as a single dose injection.
  Other Names: Naropin; Toradol; Sprix; Acuvail; Acular; EpiPen; Adrenaclick; Medihaler-Epi; Twinject; Kapvay; Catapres; Duraclon; Nexiclon
  Arms: Randomized Group A [Cocktail Injection]; Randomized Group B [Cocktail Injection Plus Exparel]
Drug: Exparel — Administered 20 minutes+ before additional medications.
  Other Names: Bupivacaine Liposome
  Arms: Randomized Group B [Cocktail Injection Plus Exparel]; Randomized Group C [Marcaine Plus Exparel]
Drug: Marcaine — Administered 20 minutes or more after Exparel is administered.
  Other Names: Bupivacaine Hydrochloride; Bupivacaine
  Arms: Randomized Group C [Marcaine Plus Exparel]

SUMMARY:
A prospective, randomized control study will be conducted to compare postoperative pain control in a series of patients treated with either:

1. a local cocktail.
2. a local cocktail plus Exparel.
3. marcaine plus Exparel prior to wound closure following knee arthroplasty.

DETAILED DESCRIPTION:
As an alternative to the various injection cocktails, Exparel, a liposomal-coated bupivicaine, was introduced as a long-acting form of bupivicaine, a local anesthetic. This new technology has been utilized by numerous orthopedic joint surgeons. Since its introduction there have been studies showing varying results in terms of postoperative pain control.

Therefore, it is our purpose to conduct a prospective, randomized control study to compare postoperative pain control in a series of patients treated with either:

1. a local cocktail.
2. a local cocktail plus Exparel.
3. marcaine plus Exparel prior to wound closure following knee arthroplasty.

METHODOLOGY

Subjects will be randomized preoperatively into three different groups on total knee subjects done at three different facilities. This study is single blinded study. The visual pain scale from 1-10 will be used to determine pain control at 3, 12, 24, and 48 hour time intervals postoperatively. Postoperative narcotic use will also be monitored at the same time intervals.

ELIGIBILITY:
Inclusion Criteria:

* Institutional Review Board (IRB) review has been conducted and approval of the study has been obtained
* The subject underwent a primary total knee replacement under adductor canal block with general anesthesia

Exclusion Criteria:

* The subject is a minor
* The subject is on chronic narcotics
* The subject has an indwelling pain pump
* The subject is having a knee revision surgery
* The subject is having a partial knee replacement
* The subject has a history of sepsis in a previously replaced joint
* The subject has back pain
* The subject has radicular pain
* The subject suffers from depression
* The subject has fibromyalgia
* The subject is currently involved in any personal injury litigation, medical-legal, or worker's compensation claims

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The visual pain scale from 1-10 will be used to determine changes in pain control at 3, 12, 24, and 48 hour time intervals postoperatively. | Pain control intervals will be assessed at 3, 12, 24, and 48 hour time intervals postoperatively.